CLINICAL TRIAL: NCT06395116
Title: "Influence of Fabrication Technique on Microbial Adhesion and Biofilm Formation to Conventional, Milled, and 3D-Printed Resin Denture Base Materials
Brief Title: Microbial Adhesion and Biofilm Formation on Denture Base Materials
Status: Active, not recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Tanta University (Other); Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mohammed Elsawy, lecturer, Department of prosthodontics, principle investigator, Menoufia University
Other Study IDs: R-RP-1-24-3091
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Response; Microbial Colonization; Denture Stomatitis
Keywords: Microbial adhesion, Biofilm formation, Denture base
MeSH Terms: conditions — Communicable Diseases; Stomatitis, Denture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventionl self cure acrylic group: Constructed from heat cured acrylic resin
  Interventions: Other: Denture base material
- 3D printed acrylis resin group: Manufactured by additive manufacturing technique
  Interventions: Other: Denture base material
- Milled acrylic resin group: Manufactured by milled technique
  Interventions: Other: Denture base material

INTERVENTIONS:
Other: Denture base material — Denture base material constructed with different techniques for completely edentulous populations

SUMMARY:
Polymethylmethacrylate (PMMA) has been the material of choice for fabricating complete dentures for more than 80 years now.(1,2) As a material it is easy to handle and can be easily repaired and polished. PMMA while being a low-cost material has good esthetics. Some disadvantages of PMMA as a material are surface roughness and porosities which lead to staining, plaque accumulation and bacterial adhesion over time.

Among the various factors that can influence microbial attachment to surfaces, surface roughness, hydrophilicity and free surface energy of PMMA are most important. Carboxylate and methyl ester groups found in PMMA make it a very hydrophilic material with a large amount of free surface energy. Despite the influence of the chemical composition, processing methods play the most important role in developing surface roughness.

DETAILED DESCRIPTION:
PMMA for dentures may be processed by conventional techniques like compression moulding or injection moulding with the conventional pack and press technique being considered the 'gold standard' when it comes to processing methods as it has successfully withstood the test of time. With the advent of technology CAD/CAM milling is now being used to mill dentures from pre-polymerized blocks of acrylic resin. At the same time 3D printing/Rapid prototyping technology is also being used to print denture bases with acrylic resins. Both these technologies eliminate the need for conventional flasking and processing methods. The rapid prototyping technique involves serial apposition of resin layers on a custom designed support structure. These layers are hardened by curing with either visible light, UV Light, heat or laser depending upon the technique used. This process is repeated until the designed structure is completely formed. The milling or subtractive technique on the other hand uses pre-polymerized commercially manufactured PMMA blanks (Pucks) which are made under high pressure. This technique allows for the material to have superior mechanical properties.

In reviewing the literature, no clinical studies were performed to compare which method of PMMA denture construction can reduce the amount of microbial colonization while there are a lot of invitro studies was performed.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous populations.
* Good physical and mental health.
* No systemic disease

Exclusion Criteria:

* Partially edentulous populations.
* Patients with smoking more than 10 citrates day.
* Patients with systemic diseases.
* Patients undergrown radiotherapy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Completely edentulous population who attended at the faculty of Dentistry, Menoufia University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Biofilm formation | 3 years
  such as Candida Albian's and Staphylococcus Aureus colonies per ml

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. El-Sawy, PhD, Study Director — Menoufia University
Locations (1):
- Mohammed A. El-Sawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
Only with permission from the corresponding author